CLINICAL TRIAL: NCT00270556
Title: Phase II, Open-Label,Randomised, Comparator Study of Substitution w/Tenofovir or Abacavir in HIV-1 Infected Individuals, w/Viral Load Less 50 Copies/mL, Receiving a Thymidine Analogue (Zidovudine or Stavudine) as Part of HAART.
Brief Title: Phase II Comparator Study of Substitution of Tenofovir or Abacavir Receiving Thymidine Analogue as Part of HAART.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Other Study IDs: GS-02-1008
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: HIV
Keywords: Treatment Experienced
MeSH Terms: interventions — Tenofovir; abacavir

INTERVENTIONS:
Drug: tenofovir disoproxil fumarate
Drug: Abacavir

SUMMARY:
This 48 week study is designed to compare the substitution of the thymidine analogues zidovudine (ZDV) or stavudine (D4T) with either tenofovir DF or abacavir, in patients treated with highly active antiretroviral therapy (HAART), and show improved outcomes on total limb fat mass, improved body shape by dual energy x-ray absorptiometry (DEXA) and computed tomography (CT) scans and improved cholesterol and tryglicerides.

DETAILED DESCRIPTION:
A previous study substituting zidovudine or stavudine to abacavir in patients with severe or moderate lipoatrophy has shown an increase in limb fat (DEXA). This study was conducted over a 24 week period and although improved outcomes were documented by objective measures, DEXA scans, subjective observation did not correspond. Longer-term follow up of these patients is required.

This 48 week study is designed to compare the substitution of the thymidine analogues zidovudine (ZDV) or stavudine (D4T) with either tenofovir DF or abacavir, in patients treated with highly active antiretroviral therapy (HAART), and show improved outcomes on total limb fat mass, improved body shape by dual energy x-ray absorptiometry (DEXA) and computed tomography (CT) scans and improved cholesterol and tryglicerides.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are male or female less than or equal to 18 years of age. HIV-1 infected as documented by a licensed HIV-1 antibody ELISA. Female subjects of childbearing potential must have a negative serum pregnancy test (beta-HCG) within 28 days of trial day 1. Women of childbearing potential must agree to use a barrier method of contraception. Female subjects must not be pregnant or lactating. Able to understand and provide written informed consent in the opinion of the investigator. Subjects have clinical lipoatrophy at greater then or equal to 1 body/facial site in the investigator's opinion. Subjects currently receiving nucleoside analogue regimen including stavudine (d4T) or zidovudine (ZDV). Subjects who are stable on current therapy for greater than or equal to 16 weeks. Subjects with no prior exposure to tenofovir, abacavir or adefovir. Subjects with no known K65R, 69S mutations or 3 or more thymidine analogue mutations. Subjects with documented viral load less than 50 copies/mL on 2 consecutive occasions including most recent clinic attendance.

Exclusion Criteria:

* Subjects who are unlikely to complete the 48 week trial period. Currently active opportunistic disease or documented wasting syndrome. Currently receiving chemotherapy for malignancy. Subjects who are unlikely to retain viral response after switching based on treatment or transmission history. Currently receiving an insulin sensitising agent (glitazone or metformin). Anabolic steriods in the last 16 weeks other than testosterone at replacement doses (less than or equal to 250 mg/2 weekly). Growth hormone use in the last 16 weeks. Statin therapy (HMG CoA reductase inhibitor) commenced in the last 16 weeks (patients stable on statins may be included). Current alcohol or illicit drug use which may interfer with the subjects ability to comply with the dosing schedule and protocol evaluations. Receiving concurrent medications that in the opinion of the investigator and according to drug product labeling will result in clinically significant interactions with tenofovir or abacavir. Pregnant or breast feeding. Previously received more than 3 months zidovudine monotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Avila, MD, Study Director — Gilead Sciences

REFERENCES:
- See also: Gilead website — http://www.Gilead.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-02-1008_synopsis.pdf